CLINICAL TRIAL: NCT00001262
Title: Early Copper Histidine Therapy in Menkes Disease
Brief Title: Copper Histidine Therapy for Menkes Diseases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 900149; 90-CH-0149
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-09

CONDITIONS: Kinky Hair Syndrome
Keywords: Menkes; Copper; X-Linked; Neurodegeneration; ATP7A
MeSH Terms: conditions — Menkes Kinky Hair Syndrome; Nerve Degeneration | interventions — copper histidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Copper histidine (Experimental)
  Interventions: Drug: Copper Histidine

INTERVENTIONS:
Drug: Copper Histidine

SUMMARY:
Menkes Disease is a genetic disorder affecting the metabolism of copper. Patient with this disease are both physically and mentally retarded. Menkes disease is usually first detected in the first 2-3 months of life. Infant males born with the disease fail to thrive, experience hypothermia, have delayed development, and experience seizures. These infants also have characteristic physical features such as changes of their hair and face. Females may also have changes in hair and skin color, but rarely have significant medical problems.

Appropriate treatment of Menkes Disease requires that the disease be diagnosed early and treatment started before irreversible brain damage occurs. The aim of treatment is to bypass the normal route of absorption of copper through the gastrointestinal tract. Copper must then be delivered to brain cells and be available for use by enzymes.

Copper histidine is a copper replacement that can be injected directly into the body to avoid absorption through the gastrointestinal tract. However, studies have shown the genetic abnormalities causing Menkes disease cannot simply be corrected by copper replacement injections.

The genetic abnormality causing Menkes disease can vary in its severity. Patients with a genetic abnormality that may still permit some production of the enzymes required to process copper may receive benefit from early treatment with copper replacement. However, patients with severe abnormalities of the genes responsible for copper metabolism may receive no benefit from copper replacement.

The purpose of this study is to continue to evaluate the effects of early copper histidine in Menkes disease patients and to correlate specific molecular defects with responses to treatment.

DETAILED DESCRIPTION:
Menkes disease is an X-linked recessive neurodegenerative disorder caused by defects in a gene that encodes an evolutionarily conserved copper-transporting ATPase (ATP7A). Several issues must be addressed in configuring therapeutic strategies for this disorder: (a) affected infants must be identified and treatment commenced very early in life before irreparable neurodegeneration occurs, (b) the block in intestinal absorption of copper must be bypassed, (c) circulating copper must be delivered to the brain, and (d) copper must be available to enzymes within cells that require it as a cofactor.

Very early, pre-symptomatic therapy with copper injections has been associated with improved overall survival and, in some patients - based on their molecular defects, with vastly better neurological outcomes in comparison to the usual natural history of this disorder. The purpose of this study is to continue to provide early copper treatment to other newborn infants diagnosed as having Menkes disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Newborn infants in whom Menkes disease is confirmed on biochemical or molecular grounds and in whom no neurological symptoms are present are eligible for enrollment in this study.

EXCLUSION CRITERIA:

Newly identified patients classified as symptomatic at the time of diagnosis, and affected individuals with mild phenotypes are not currently eligible for this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1990-06; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Kaler, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Kaler SG, Buist NR, Holmes CS, Goldstein DS, Miller RC, Gahl WA. Early copper therapy in classic Menkes disease patients with a novel splicing mutation. Ann Neurol. 1995 Dec;38(6):921-8. doi: 10.1002/ana.410380613. PMID 8526465
- [Result] Kaler SG, Holmes CS, Goldstein DS, Tang J, Godwin SC, Donsante A, Liew CJ, Sato S, Patronas N. Neonatal diagnosis and treatment of Menkes disease. N Engl J Med. 2008 Feb 7;358(6):605-14. doi: 10.1056/NEJMoa070613. PMID 18256395
- [Result] Kaler SG, Gahl WA, Berry SA, Holmes CS, Goldstein DS. Predictive value of plasma catecholamine levels in neonatal detection of Menkes disease. J Inherit Metab Dis. 1993;16(5):907-8. doi: 10.1007/BF00714295. No abstract available. PMID 8295415
- [Result] Kaler SG, Westman JA, Bernes SM, Elsayed AM, Bowe CM, Freeman KL, Wu CD, Wallach MT. Gastrointestinal hemorrhage associated with gastric polyps in Menkes disease. J Pediatr. 1993 Jan;122(1):93-5. doi: 10.1016/s0022-3476(05)83496-1. PMID 8419622
- [Result] Grange DK, Kaler SG, Albers GM, Petterchak JA, Thorpe CM, DeMello DE. Severe bilateral panlobular emphysema and pulmonary arterial hypoplasia: unusual manifestations of Menkes disease. Am J Med Genet A. 2005 Dec 1;139A(2):151-5. doi: 10.1002/ajmg.a.31001. PMID 16278898
- [Result] Price DJ, Ravindranath T, Kaler SG. Internal jugular phlebectasia in Menkes disease. Int J Pediatr Otorhinolaryngol. 2007 Jul;71(7):1145-8. doi: 10.1016/j.ijporl.2007.02.021. Epub 2007 May 4. PMID 17482283
- [Result] Hicks JD, Donsante A, Pierson TM, Gillespie MJ, Chou DE, Kaler SG. Increased frequency of congenital heart defects in Menkes disease. Clin Dysmorphol. 2012 Apr;21(2):59-63. doi: 10.1097/MCD.0b013e32834ea52b. PMID 22134099
- [Result] Kaler SG, Gallo LK, Proud VK, Percy AK, Mark Y, Segal NA, Goldstein DS, Holmes CS, Gahl WA. Occipital horn syndrome and a mild Menkes phenotype associated with splice site mutations at the MNK locus. Nat Genet. 1994 Oct;8(2):195-202. doi: 10.1038/ng1094-195. PMID 7842019
- [Result] Liu PC, Chen YW, Centeno JA, Quezado M, Lem K, Kaler SG. Downregulation of myelination, energy, and translational genes in Menkes disease brain. Mol Genet Metab. 2005 Aug;85(4):291-300. doi: 10.1016/j.ymgme.2005.04.007. PMID 15923132
- [Result] Kaler SG, Das S, Levinson B, Goldstein DS, Holmes CS, Patronas NJ, Packman S, Gahl WA. Successful early copper therapy in Menkes disease associated with a mutant transcript containing a small In-frame deletion. Biochem Mol Med. 1996 Feb;57(1):37-46. doi: 10.1006/bmme.1996.0007. PMID 8812725
- [Result] Tang J, Donsante A, Desai V, Patronas N, Kaler SG. Clinical outcomes in Menkes disease patients with a copper-responsive ATP7A mutation, G727R. Mol Genet Metab. 2008 Nov;95(3):174-81. doi: 10.1016/j.ymgme.2008.06.015. Epub 2008 Aug 26. PMID 18752978
- [Result] Kaler SG, Tang J, Donsante A, Kaneski CR. Translational read-through of a nonsense mutation in ATP7A impacts treatment outcome in Menkes disease. Ann Neurol. 2009 Jan;65(1):108-13. doi: 10.1002/ana.21576. PMID 19194885
- [Result] Kaler SG, Liew CJ, Donsante A, Hicks JD, Sato S, Greenfield JC. Molecular correlates of epilepsy in early diagnosed and treated Menkes disease. J Inherit Metab Dis. 2010 Oct;33(5):583-9. doi: 10.1007/s10545-010-9118-2. Epub 2010 Jul 21. PMID 20652413
- [Result] Desai V, Donsante A, Swoboda KJ, Martensen M, Thompson J, Kaler SG. Favorably skewed X-inactivation accounts for neurological sparing in female carriers of Menkes disease. Clin Genet. 2011 Feb;79(2):176-82. doi: 10.1111/j.1399-0004.2010.01451.x. PMID 20497190
- [Result] Kaler SG. Neurodevelopment and brain growth in classic Menkes disease is influenced by age and symptomatology at initiation of copper treatment. J Trace Elem Med Biol. 2014 Oct;28(4):427-30. doi: 10.1016/j.jtemb.2014.08.008. Epub 2014 Aug 28. PMID 25281031
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1990-CH-0149.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Early: Classic Menkes disease: Copper histidine treatment beginning within 1 month of age
- Late: Classic Menkes disease: Copper histidine treatment beginning after 1 month of age and after onset of symptoms
- Mild: Milder variants of Menkes disease: Copper histidine treatment beginning late (L) and after onset of (milder) symptoms
Period: Overall Study
Arm/Group | Early | Late | Mild
Started | 35 | 22 | 3
Completed | 25 | 8 | 3
Not Completed | 10 | 14 | 0
Not completed — Death | 10 | 11 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early | Late | Mild | Total
Number analyzed (Participants) | 35 | 22 | 3 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 22 | 3 | 60
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 34 | 22 | 3 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 30 | 21 | 3 | 54
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 1 | 0 | 10
  White | 22 | 19 | 3 | 44
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Gross Motor Development at 36 Mos of Age or at Death (Mos)
Description: This was measured based on the Denver Developmental Screening Test (DDST) I or II for age-appropriate gross motor development in apparently normal healthy subjects at specific ages (in months). The DDST employs a grid to assess expected developmental milestones in relation to chronologic age.
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - months
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - months | 13.743 (12.200) | 2.455 (2.154) | 15.667 (9.815)

2. Primary Outcome: Fine Motor Adaptive Development at 36 Mos of Age or at Death (Mos)
Description: This was measured based on the Denver Developmental Screening Test (DDST) I or II for age-appropriate fine motor development in apparently normal healthy subjects at specific ages (in months). The DDST employs a grid to assess expected developmental milestones in relation to chronologic age.
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - Months
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - Months | 16.200 (12.762) | 2.409 (1.652) | 17.667 (13.204)

3. Primary Outcome: Personal-Social Development at 36 Mos of Age or at Death (Mos)
Description: This was measured based on the Denver Developmental Screening Test (DDST) I or II for age-appropriate personal-social development in apparently normal healthy subjects at specific ages (in months). The DDST employs a grid to assess expected developmental milestones in relation to chronologic age.
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - Months
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - Months | 17.657 (13.482) | 3.364 (3.499) | 17.667 (15.308)

4. Primary Outcome: Language Development at 36 Mos of Age or at Death (Mos)
Description: This was measured based on the Denver Developmental Screening Test (DDST) I or II for age-appropriate language development in apparently normal healthy subjects at specific ages (in months). The DDST employs a grid to assess expected developmental milestones in relation to chronologic age.
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - Months
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - Months | 15.800 (12.034) | 3.227 (2.943) | 21.000 (9.539)

5. Secondary Outcome: Somatic Growth Percentiles at 3 Years of Age (or at Age of Death) - Weight Percentile
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - Percentile
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - Percentile | 12.086 (19.589) | 11.273 (17.097) | 5.000 (8.660)

6. Secondary Outcome: Somatic Growth Percentiles at 3 Years of Age (or at Age of Death) - Length Percentile
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - Percentile
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - Percentile | 8.286 (13.501) | 15.455 (23.192) | 28.333 (40.723)

7. Secondary Outcome: Somatic Growth Percentiles at 3 Years of Age (or at Age of Death) - Head Circumference Percentile
Time Frame: 36 months or death
Measure: Mean (Standard Deviation); unit: Other - Percentile
Arm/Group | Early | Late | Mild
Number analyzed (Participants) | 35 | 22 | 3
Other - Percentile | 33.286 (27.060) | 11.136 (14.551) | 18.333 (27.538)

ADVERSE EVENTS:
Time Frame: 36 months or death
Arm/Group | Early | Late | Mild
Serious Adverse Events (participants affected / at risk) | 10/35 | 11/22 | 0/3
Other Adverse Events (participants affected / at risk) | 0/35 | 0/22 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early (N=35) | Late (N=22) | Mild (N=3)
Death (Nervous system disorders) | 10 (10) | 11 (11) | 0 (0) — Menkes disease
Dehydration (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No